CLINICAL TRIAL: NCT01904357
Title: USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System in Pediatric Subjects of 10-12 Years (Inclusive) Scheduled for Surgery
Brief Title: Pediatric Cefazolin PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: B. Braun Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HC-G-H-1202
Record Dates: First submitted 2013-07-15; First posted 2013-07-22 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Infections
Keywords: Cefazolin, Pediatric
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefazolin 1 GM Injection (Active Comparator): Subjects weighing ≥25 kg and < 50 kg will receive the 1g dose.
  Interventions: Drug: Cefazolin 1 GM Injection
- Cefazolin 2 GM Injection (Active Comparator): Subjects weighing ≥50 kg to ≤85 kg will receive the 2g dose.
  Interventions: Drug: Cefazolin 2 GM Injection

INTERVENTIONS:
Drug: Cefazolin 1 GM Injection — Subjects weighing ≥25 kg and < 50 kg will receive the 1g dose.
  Arms: Cefazolin 1 GM Injection
Drug: Cefazolin 2 GM Injection — Subjects weighing ≥50 kg to ≤85 kg will receive the 2g dose.
  Arms: Cefazolin 2 GM Injection

SUMMARY:
The primary objective of this study is:

• To examine the pharmacokinetics (PK) of cefazolin in children aged 10 to 12 years (inclusive) receiving weight-dependent 1gram (g) or 2g of cefazolin intravenous (IV) delivered over 30 minutes via the DUPLEX® drug delivery system for surgical prophylaxis.

The secondary objectives of this study are:

* To compare the PK data in children aged 10 to 12 years (inclusive)receiving 1g or 2g of cefazolin IV delivered over 30 minutes via the DUPLEX® drug delivery system with modeling data for adolescents aged 13-17 years (inclusive) and historical data from adults receiving a single 2g dose of cefazolin.
* To assess the safety of a single dose of cefazolin in children aged 10 to 12 years (inclusive) receiving 1g or 2g of cefazolin IV delivered over 30 minutes via the DUPLEX® drug delivery system for surgical prophylaxis.

DETAILED DESCRIPTION:
This is a multiple-center, open-label, PK study of cefazolin in children aged 10 to 12 years (inclusive) receiving 1g or 2 g of cefazolin delivered via the DUPLEX® drug delivery system for surgical prophylaxis. Surgery should be expected to last no longer than 3 hours. If a second dose of cefazolin is required, the subject will be excluded from the PK analysis and additional subjects will be enrolled if necessary to obtain eight evaluable subjects. The surgical procedures may be performed in an outpatient or inpatient setting but subjects must be available to complete the planned 8-hour PK sampling as noted below. Study drug will be administered by continuous infusion over a 30-minute period using an infusion pump. Based on weight at Day 1(Day of Surgery) (unless a weight assessment was obtained within the previous seven days that by physician judgment is felt to represent a stable weight and not have the potential to change such that the subject dose may be affected). Subjects weighing ≥25 kg and < 50 kg will receive the 1g dose. Subjects weighing ≥ 50 kg and ≤ 85 kg will receive the 2g dose. Dose groups will not be balanced by age or gender. The weight-based dosage regimen that will be employed for this study has been selected to assure that subjects will receive a dose between 20 and 40 mg/kg body weight, based on Monte Carlo simulations using adult PK data, which is consistent with current practice. Blood samples for determination of PK of cefazolin will be drawn at the following times: 15 minutes before the start of infusion (baseline), at the end of infusion, 15 and 30 minutes and 1 hour, 2 hours, 3 hours, 6 hours, and 8 hours after the end of the infusion for a total of nine blood samples. Safety will be assessed by monitoring adverse and serious adverse events based on patient history, vital signs, and physical examination. Follow-up phone calls will be placed to each subject one week post treatment to assess adverse events (AEs) and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects of 10 to 12 years (inclusive) at the time of screening and who are scheduled for any type of surgery requiring single-dose perioperative cefazolin prophylaxis
2. The subject and the subject's Legal Authorized Representative (LAR) voluntarily agree that the subject will participate in this study and the LAR signs an Institutional Review Board-approved informed consent and Health Insurance Portability and Accountability Act Authorization prior to the performance of any of the screening procedures

Exclusion Criteria:

1. Known allergy or hypersensitivity to beta-lactam/cephalosporin antibiotics, corn or dextrose- containing products or solutions or any of the other ingredients of the Investigational Product (IP)
2. Pregnant or nursing females
3. Subjects with impaired renal function based on the Revised Schwartz Formula using actual body height, i.e., estimated creatinine clearance ≤ 80 mL/minute/1.73m2 (performed at Screening only if test results are not available within 3 months prior to the planned surgical procedure); the Schwartz GFR is:

   * GFR = 0.41 x height (cm)
   * Serum creatinine (mg/dL)
4. Have surgery scheduled and planned to last > 3 hours
5. Body Weight <25.0 kg or > 85.0 kg
6. Other laboratory tests, obtained as standard of care, that are outside the normal limits according to site's laboratory reference ranges or are considered by the Investigator, to be clinically significant
7. Administration of cefazolin within the past seven days
8. Administration of any medication (e. g., prescription, herbal, over-the-counter medication(s) or dietary supplements) or medication known to interact with the cefazolin that might interfere with the study drug or study procedures
9. Prior medical history of human immunodeficiency virus, hepatitis C virus, or hepatitis B virus
10. Alcohol abuse or drug abuse
11. Received an investigational drug/device within 30 days of the first dose of study drug
12. Clinically relevant medical condition(s) likely to interfere with the evaluation of the trial drug (e.g., pulmonary disease, metabolic disorders, active malignant disease, autoimmune diseases, and cardiovascular disease)
13. Any planned medical intervention or personal event that might interfere with the ability to comply with the study requirements
14. Any condition (s) that in the opinion of the PI would compromise the safety of the subject or the quality of the data
15. Unable or unwilling to adhere to the study-specified procedures and restrictions

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Single dose study to evaluate the pharmacokinetics of Cefazolin for Injection USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System in pediatric subjects of 10-12 years (inclusive) scheduled for surgery | 8 hours
  To examine the pharmacokinetics (PK) of cefazolin in children aged 10 to 12 years (inclusive) receiving weight-dependent 1gram (g) or 2g of cefazolin intravenous (IV) delivered over 30 minutes via the DUPLEX® drug delivery system for surgical prophylaxis.

SECONDARY OUTCOMES:
Single dose study to evaluate the pharmacokinetics of Cefazolin for Injection USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System in pediatric subjects of 10-12 years (inclusive) scheduled for surgery | 8 Days
  To compare the PK data in children aged 10 to 12 years (inclusive)receiving 1g or 2g of cefazolin IV delivered over 30 minutes via the DUPLEX® drug delivery system with modeling data for adolescents aged 13-17 years (inclusive) and historical data from adults receiving a single 2g dose of cefazolin.
  •
Safety of Cefazolin Dose of 1g or 2 g in children aged 10-12 years of age | 8 days
  To assess the safety of a single dose of cefazolin in children aged 10 to 12 years (inclusive) receiving 1g or 2g of cefazolin IV delivered over 30 minutes via the DUPLEX® drug delivery system for surgical prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Schmitz, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (2):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Toledo Children's Hospital, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nahata MC, Durrell DE, Ginn-Pease ME, King DR. Pharmacokinetics and tissue concentrations of cefazolin in pediatric patients undergoing gastrointestinal surgery. Eur J Drug Metab Pharmacokinet. 1991 Jan-Mar;16(1):49-52. doi: 10.1007/BF03189874. PMID 1936061
- [Derived] Schmitz ML, Blumer JL, Cetnarowski W, Rubino CM. Determination of appropriate weight-based cutoffs for empiric cefazolin dosing using data from a phase 1 pharmacokinetics and safety study of cefazolin administered for surgical prophylaxis in pediatric patients aged 10 to 12 years. Antimicrob Agents Chemother. 2015 Jul;59(7):4173-80. doi: 10.1128/AAC.00082-15. Epub 2015 May 4. PMID 25941220